CLINICAL TRIAL: NCT03981809
Title: Development and Validation of a Screening Tool to Identify the Dominant Pain Mechanism in Cancer Survivors With Persistent Pain
Brief Title: Screening Tool to Identify the Dominant Pain Mechanism in Cancer Survivors: PainsCan
Acronym: PainsCan
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, An De Groef, Principal investigator An De Groef, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62584
Record Dates: First submitted 2019-05-20; First posted 2019-06-11 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cancer Survivors; Cancer Pain
Keywords: Pain; Cancer; Chronic pain; Persistent pain
MeSH Terms: conditions — Cancer Pain; Pain; Neoplasms; Chronic Pain | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic test ("PainsCan") for the identification of the dominant pain mechanisms in cancer survivers with persistent pain — Easy-to-use screening tool to identify the dominant pain mechanism by using quick clinical tests and compare their accuracy and validity with complicated reference tests.

SUMMARY:
Development and internal validation of an easy-to-use tool for clinical pain assessment. The tool has to be applicable in any clinical practice and without the need for expensive and complicated hospital tools to identify the source of persistent pain after the treatment of cancer.

DETAILED DESCRIPTION:
An adequate selection of physiotherapy treatment for persistent pain after the treatment of cancer, depends highly on the mechanism of the pain.

Pain can arise from a damaged nerve or tissue (skin, lymphatic system...). But when pain becomes chronic, alterations to the central nervous system can occur, as regulations of the facilitating and inhibiting mechanisms. These alterations may cause central sensitization pain. The body is now sensitized and cannot distinct harmful from harmless stimuli.

Each type of pain requires a specific treatment, therefore identification of the pain mechanism is crucial. Up till now, expensive and complex tests were performed in a hospital setting to determine if a patient suffers from neuropathic, nociceptive or central sensitization pain. This study aims for developping an assessment tool that does not require expensive devices but can be easily performed by any physiotherapist, within the timeframe of a standard consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for primary cancer: breast, prostate, lung/bronchus, colon/rectum, gynecologic (uterus or ovary)
* Complete remission
* Curative treatment finished
* Ongoing hormonal and targeted treatment permitted
* Patient experiences pain (NRS minimum 3/10 during the past week)

Exclusion Criteria:

* Active metastasis
* Palliative status
* Other type of cancer than mentioned in inclusion criteria
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients older than 18, in complete remission, who experience pain scored with a minimum of 3/10 (0 being no pain at all and 10 being the worst pain imaginable). The patients do not have metastasis and are not in a palliative status, nor are they pregnant or diagnosed with a cancer type other than breast, prostate, lung/bronchus, colon/rectum or gynecologic cancer.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Douleur Neuropathic 4 questions (DN4) questionnaire | 2 minutes
  Neuropathic pain: pain that arises from a damaged nerve is assessed with a questionnaire (1)
Quantitative sensory testing | 20 minutes
  Neuropathic pain: pain that arises from a damaged nerve is assessed by measuring thermal thresholds (2)
Pain mapping | 1 minute
  Neuropathic pain: pain that arises from a damaged nerve is assessed by painting affected areas on a body chart (3)
Central Sensitization Inventory (CSI) questionnaire | 5 minutes
  Central sensitization pain: pain caused by changes in the central nervous system is assessed with a questionnaire (1)
Conditioned pain modulation | 10 minutes
  Central sensitization pain: pain caused by changes in the central nervous system is assessed with a thermal test (2)
Temporal summation | 2,5 minutes
  Central sensitization pain: pain caused by changes in the central nervous system is assessed with a series of touch stimuli (3)
Diffuse pain | 0,5 minute
  Central sensitization pain: pain caused by changes in the central nervous system is assessed by painting affected areas on a body chart (4)
Manual palpation | 3 minutes
  Central sensitization pain: pain caused by changes in the central nervous system is assessed by applying pressure with manual palpation (5)
Evaluation of skin | 20 seconds
  Nociceptive pain: pain that arises from a damaged tissue is assessed by visual evaluation of the skin condition (1)
Lymphedema | 4 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by examining the presence of lymphedema by measuring the circumference of the arm (2)
Joint pain | 30 seconds
  Nociceptive pain: pain that arises from a damaged tissue is assessed by examining if several joints are sore, especially in the morning (3)
Active mobility | 2,5 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by examining the movements the patient can perform (4)
Passive mobility | 3,5 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by examining the movements the clinician can perform on the patient (5)
Strength | 1,5 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by the strength the patient can perform in a specific movement (6)
Scar tissue | 2 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by examining the elasticity of the scar tissue by manual palpation of the clinician (7)
Axillary web syndrome | 2 minutes
  Nociceptive pain: pain that arises from a damaged tissue is assessed by visually examining the presence of lymph cords in the axilla (8)

SECONDARY OUTCOMES:
Pain catastrophizing scale | 6 minutes
  Pain catastrophizing scale
Depression, anxiety and stress | 7 minutes
  Depression Anxiety and Stress Scale (DASS-21)
Pain Self-efficacy and Expectations: questionnaire | 5 minutes
  Pain self-efficacy and expectations questionnaire
Pain character: questionnaire | 4 minutes
  McGill Pain questionnaire
Pain disability: Pain Disability Index | 3 minutes
  Pain Disability Index
Pain intensity: Visual Analogue Scale | 1 minute
  Visual Analogue Scale at the moment, worst and least pain during the past week
Pain questionnaire | 30 seconds
  Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, Prof., Study Director — UZ Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided